CLINICAL TRIAL: NCT05998421
Title: The Effects of Acupuncture on the Natural Pregnancy in Patients With Recurrent Abortion: a Randomized Prospective Trial
Brief Title: The Effects of Acupuncture on the Natural Pregnancy in Patients With Recurrent Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianmei Xia (Other)
Responsible Party: Sponsor-Investigator, Jianmei Xia, Deputy Chief Physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023003
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Acupuncture; Recurrent Spontaneous Abortion; Ultrasound Therapy; Coagulation
MeSH Terms: conditions — Abortion, Spontaneous; Thrombosis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the drug group (control group) (Active Comparator): The patients in the control group accepted routine aspirin and heparin treatment. Two months before pregnancy, 50 mg of aspirin (Chenxin Pharmaceutical, China) was taken orally once a day.
  Interventions: Drug: routine aspirin and heparin treatment
- the drug-accompanied-by-acupuncture group (acupuncture group) (Experimental): The patients in the acupuncture group accepted acupuncture treatment weekly from the second day of menstruation and three times in one cycle.
  Interventions: Procedure: acupuncture; Drug: routine aspirin and heparin treatment

INTERVENTIONS:
Procedure: acupuncture — The patients in the acupuncture group accepted acupuncture treatment weekly from the second day of menstruation and three times in one cycle. Seirin 0.2-×30-mm acupuncture needles were used. First, needles were inserted into Shenting (GV 24) and bilateral Benshen (G 13) to relieve uneasiness of mind. Then, they were inserted into Chung wan (cv 12), Qihai (CV6), Guan yuan, chung chi (cv 3), bilateral Guiai (S 29) and Zigong (Extra 16) to recuperate energy. Finally, bilateral Tsusanli (st 36), Yinlingch'uan (sp 9) and San yin chiao (sp 6) were used to soothe the liver and tonify the spleen and kidney. Each acupuncture treatment session lasted 30 minutes, with mostly bilateral needle retention over 20-30 minutes for evens techniques.
  Arms: the drug-accompanied-by-acupuncture group (acupuncture group)
Drug: routine aspirin and heparin treatment — The patients accepted routine aspirin and heparin treatment. Two months before pregnancy, 50 mg of aspirin (Chenxin Pharmaceutical, China) was taken orally once a day.

SUMMARY:
Recurrent spontaneous abortion (RSA) is a common pregnancy complication in women of reproductive age and the cause of RSA remains largely unclear. Acupuncture is widely used in clinical practice to treat infertility and abortion. The role of acupuncture in the treatment of infertility is still unclear. The investigators conducted a randomized, prospective, controlled clinical trial to investigate its potential impact on pregnancy outcome. Herein, the investigators not only evaluated the changes in patients' psychological stress before and after treatment but also followed up on pregnancy outcomes. In addition, changes in uterine artery blood flow were observed by ultrasound. Changes in coagulation-related indicators were also detected.

DETAILED DESCRIPTION:
To better illustrate the effectiveness and mechanism of acupuncture in infertility, especially in RSA patients, the investigators conducted a randomized, prospective, controlled clinical trial to investigate its potential impact on pregnancy outcome. Herein, the investigators not only evaluated the changes in patients' psychological stress before and after treatment but also followed up on pregnancy outcomes. In addition, changes in uterine artery blood flow were observed by ultrasound. Changes in coagulation-related indicators were also detected. The investigators hypothesized that acupuncture could promote and improve pregnancy by improving uterine artery blood flow and relieving patients' anxiety symptoms. To our knowledge, it has never been reported before.

ELIGIBILITY:
Inclusion Criteria:

* had a previous RSA history;
* had a normal body mass index (BMI) of 18-25 kg/m2;
* had no acute infection of the abdomen and low back skin;
* had no history of liver or kidney disease.

Exclusion Criteria:

* acute infection in the abdomen or lower back
* planning assisted reproductive technologies (ART) in the next 3 months

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
The effect of acupuncture on pregnancy outcome in patients with recurrent spontaneous abortion | average of 1 year
  The pregnancy outcome of each patient was followed-up. The outcomes of natural pregnancy include normal clinical pregnancy(intrauterine pregnancy and pregnancy week ≥28) and adverse pregnancy. The latter includes biochemical pregnancy, spontaneous abortion and ectopic gestation.
The change of blood indicators related to blood coagulation function after acupuncture1 | average of half of a year
  Changes in blood indicators related to blood coagulation function, such as platelet maximum aggregation rate (MAR, inducted by arachidonic acid (AA) and adenosine diphosphate (ADP)), were also detected before and after treatment.
The effect of acupuncture on blood flow impedance in the uterine arteries before and after each treatment cycle | average of half of a year
  Patients in both groups were scheduled for vaginal ultrasound in the mid luteal phase to monitor the blood flow impedance in the uterine arteries before and after each treatment cycle, measured as the uterine artery (UA) systolic/diastolic (S/D) blood flow ratio.
The effect of acupuncture on patients' mental anxiety status before and after each treatment cycle | average of half of a year
  Generalized anxiety disorder (GAD-7) was used to assess patients' mental anxiety status. Each item has a score of 0-3, totaling 7 items, with a total score of 0-21. The higher the score, the more severe it becomes.
The change of blood indicators related to blood coagulation function after acupuncture2 | average of half of a year
  Changes in blood indicators related to blood coagulation function, such as D-dimer (D-D)were also detected before and after treatment.
The change of blood indicators related to blood coagulation function after acupuncture3 | average of half of a year
  Changes in blood indicators related to blood coagulation function, such as prothrombin time (PT) and activated partial thromboplastin time (APTT), were also detected before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmei Xia, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Jianmei Xia, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No